CLINICAL TRIAL: NCT06115148
Title: Breath Ammonia as a Malnutrition Screening Tool
Brief Title: Breath Analysis & Malnutrition
Acronym: BAM-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Jacob T. Mey, PhD RD, Assistant Professor - Research, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PBRC 2022-059
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization scheme will be blinded to the PI and biostatistician. Due to the intervention (feeding vs fasting), the participant and other study staff cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feeding (Experimental): Participants will be instructed to consume study beverages to provide >1.2 grams of protein per kilogram bodyweight and >120% of total energy needs. Energy needs will be estimated by the Mifflin-St Jeor equation multiplied by an activity factor of 1.5. Study beverages will be a mix of meal replacement shakes e.g., Ensure (Abbott Laboratories, Chicago, IL, USA) products to accommodate protein and energy needs. Study beverages will be consumed every ~3 hours to induce a perpetually fed state. Feeding will occur during waking hours, typically between 7a-11p. Breath will be collected before, during and after the intervention.
  Interventions: Other: Feeding
- Fasting (Experimental): Participants will be instructed to consume only water during the duration of the Fasting Protocol. Regardless of the randomization sequence, participants will have consumed their last meal or study beverage by 11p the night prior. Breath will be collected before, during and after the intervention.
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Feeding — Nutrition beverages will be provided to meet the nutrient needs described in the Feeding Arm.
  Arms: Feeding
Other: Fasting — Water will be consumed as described during the Fasting Arm.
  Arms: Fasting

SUMMARY:
The purpose of this research study is to understand how breath is related to nutritional status. The procedures involved in this study include blood and breath sampling, questionnaires about health history, medications, nutritional status and diet, and a physical examination. Breath markers will be compared between individuals with and without malnutrition and be compared to indicators of malnutrition. Some individuals will undergo an interventional study involving 2 days of consuming study beverages and fasting along with providing additional breath samples to see if the breath changes in response to short-term changes in nutritional status.

DETAILED DESCRIPTION:
Research Summary: This research involves a cross-sectional study investigating whether breath molecules (in particular ammonia and nitric oxide) are related to the presence and magnitude of malnutrition as measured by the gold-standard nutrition focused physical examination (NFPE). It also involves an interventional study in a subset of cross-sectional participants looking at whether acute changes in nutritional status through anabolic feeding protocols or fasting protocols is related to short term changes in breath molecules.

Purpose of the Research: The purpose is to identify early evidence of breath biomarkers of malnutrition. It uses a combination of breath analysis and current malnutrition screening tools (questionnaires).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-95 years
2. Malnutrition group (Cross-sectional study only); not involved in intervention: Diagnosed with malnutrition (verified in medical history)

Exclusion Criteria:

1. Chronic kidney, liver or pulmonary disease
2. Anabolic steroid use other than testosterone (e.g., oxandrolone)
3. Patients judged unsuitable for enrollment by the study medical investigator
4. Pregnant women or women who are nursing
5. Unable or unwilling to consume study beverages or fast for 24 hours each arm

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Breath Ammonia | Interventional: Upon waking and after the intervention, but before bed on each of the 1-day intervention arms
  Breath ammonia (ppm)

SECONDARY OUTCOMES:
Breath volatile organic compounds | Interventional: Upon waking and after the intervention, but before bed on each of the 1-day intervention arms
  Untargeted mass spectrometry on breath volatile organic compound concentration in breath
Fractional Exhaled Nitric Oxide | Interventional: Upon waking and after the intervention, but before bed on each of the 1-day intervention arms
  Fractional exhaled nitric oxide (ppb)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Mey, PhD, RD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
External investigators may request additional data access, which will be shared according to institutional policy with appropriate data sharing agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon reasonable request.
Access Criteria: According to institutional policy.